CLINICAL TRIAL: NCT03572764
Title: A Pilot Study of CPX-351 (Vyxeos™) for Transplant Eligible, Higher Risk Patients With Myelodysplastic Syndrome
Brief Title: CPX-351 (Vyxeos™) for Transplant Eligible, Higher Risk Patients With Myelodysplastic Syndrome
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201807148
Record Dates: First submitted 2018-06-18; First posted 2018-06-28 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — CPX-351; Daunorubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CPX-351 (Experimental): * CPX-351 will be given according to the assigned dose level over a minimum of a 90-minutes via IV infusion on Days 1, 3, and 5 of the first induction
  * If the treating physician elects to perform a day 14 bone marrow biopsy then, a second induction may be considered for patients in the absence of a chemoablated, hypocellular marrow on the Day 14 bone marrow assessment, if the patient has failed to achieve a marrow CR, and it is deemed safe to administer by the treating physician. The second induction uses a modified schedule in which CPX-351 will be given according to the assigned dose level on Days 1 and 3
  * In the absence of disease progression or unacceptable toxicity, the patient may continue to consolidation at the discretion of the treating physician or the patient may proceed to alloHCT after induction at the discretion of the treating physician
  Interventions: Drug: CPX-351; Procedure: Research skin biopsy; Procedure: Research blood draw; Procedure: Research bone marrow aspirate

INTERVENTIONS:
Drug: CPX-351 — -CPX-351 will be provided by Jazz Pharmaceuticals
  Other Names: Vyxeos™; Daunorubicin and cytarabine
Procedure: Research skin biopsy — -And/or buccal swab
  * Pre-treatment
  * Post-induction (no earlier than Day 28 and no later than Day 56 from last induction)
Procedure: Research blood draw — * Pre-treatment
  * Post-induction (no earlier than Day 28 and no later than Day 56 from last induction)
  * Post-consolidation 1 (if applicable)
  * Post-consolidation 2 (if applicable)
  * Post-transplant Day 30 (if applicable)
  * Post-transplant Day 100 (if applicable)
Procedure: Research bone marrow aspirate — * Pre-treatment
  * Post-induction (no earlier than Day 28 and no later than Day 56 from last induction)
  * Post-consolidation 1 (if applicable)
  * Post-consolidation 2 (if applicable)
  * Post-transplant Day 30 (if applicable)
  * Post-transplant Day 100 (if applicable)

SUMMARY:
This is a pilot and feasibility study of transplant eligible, higher risk myelodysplastic syndrome (MDS) patients to determine the safety and tolerability of a lower -dose and higher-dose CPX-351 regimen, with secondary objectives including complete remission (CR) rates and proportion of patients proceeding to transplant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myelodysplastic syndrome (MDS) with an IPSS-R score of Intermediate, High or Very High (see Appendix A) AND ≥ 5% myeloblasts in the bone marrow.
* Age 18-70 years.
* ECOG performance status ≤ 2 (see Appendix B)

Adequate renal and hepatic function as defined below:

*Total bilirubin ≤ 2.0 x IULN*

* AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
* Serum creatinine ≤ 2.0 mg/dL
* Note: If, in the opinition of the treatment physician, the bilirubin is elevated secondary to hemolysis or Gilbert's disease, the patient may be eligible after discussion with the Washington University PI.

  * Left ventricular cardiac ejection fraction ≥ 50% by echocardiography or MUGA.
  * Deemed by the treating physician to be a suitable candidate for cytotoxic induction therapy and an alloHCT candidate at the time of enrollment.
  * Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and continuing until 30 days after the last study treatment.
  * Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior treatment for MDS with disease-modifying therapy (conventional or investigational) (i.e. hypomethylator therapy, lenalidomide, or prior AML-like induction therapy intended for the therapy of MDS). Use of prior growth factor and ESA support is permitted.
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to CPX-351 or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* History of Wilson's disease or other copper-metabolism disorder.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Known active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible. Patients who are seropositive for HCV but have a negative viral load are also eligible provided that the patient has completed a course of therapy for HCV.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2021-11-27 (Actual); Study Completion 2027-03-25 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of a CPX-351 regimen in a transplant eligible, higher risk MDS population as measured by the proportion of participants who experience an adverse event by patient, type of event, and grade of event | Through 56 days after the last dose

SECONDARY OUTCOMES:
Overall response rate in MDS patients treated with CPX-351 | 56 days after the last dose
  * Overall response rate = complete remission + marrow complete remission + partial response + hematologic improvement
  * Patients will be assessed for response according to modified International Working Group (IWG) criteria for MDS
Best overall response in MDS patients treated with CPX-351 | 56 days after the last dose
  -Patients will be assessed for response according to modified International Working Group (IWG) criteria for MDS
Remission duration in MDS patients treated with CPX-351 | Through 5 years
  * Defined as the interval from the date complete remission is documented to the date of recurrence. This is determined only for patients achieving a complete remission.
  * Patients will be assessed for response according to modified International Working Group (IWG) criteria for MDS
Relapse-free survival in MDS patients treated with CPX-351 | Through 5 years
  -Patients will be assessed for response according to modified International Working Group (IWG) criteria for MDS
Progression-free survival in MDS patients treated with CPX-351 | Through 5 years
  * Defined as the interval from the date of first dose of study drug to disease progression or death from MDS.
  * Patients will be assessed for response according to modified International Working Group (IWG) criteria for MDS
Overall survival in MDS patients treated with CPX-351 | Through 5 years
  -Defined as the date of first dose of study drug to the date of death from any cause.
Complete remission + marrow complete remission rates in patients treated with CPX-351 | 56 days after the last dose
  -Patients will be assessed for response according to modified International Working Group (IWG) criteria for MDS
Post-induction mortality in MDS patients treated with CPX-351 | Day 30
  -Rate of death
Post-induction mortality in MDS patients treated with CPX-351 | Day 60
  -Rate of death
Safety and feasibility of CPX-351 consolidation therapy in MDS patients as measured by the proportion of patients who experience an adverse event by patient, type of event, and grade of event | Through 56 days after the last dose
Proportion of MDS patients treated with CPX-351 proceeding to allogeneic hematopoietic cell transplant | Through 56 days after the last dose
Overall survival in MDS patients treated with CPX-351 in patients undergoing allogeneic hematopoietic cell transplant | Day 100
  -Defined as the date of first dose of study drug to the date of death from any cause.
Overall survival in MDS patients treated with CPX-351 in patients undergoing allogeneic hematopoietic cell transplant | 1 year
  -Defined as the date of first dose of study drug to the date of death from any cause.
Non-relapse mortality in MDS patients treated with CPX-351 in patients undergoing allogeneic hematopoietic cell transplant | Day 100
Non-relapse mortality in MDS patients treated with CPX-351 in patients undergoing allogeneic hematopoietic cell transplant | 1 year
Event-free survival in MDS patients treated with CPX-351 in patients undergoing allogeneic hematopoietic cell transplant | Day 100
  * Defined as the interval from the date of first dose of study drug to date of treatment failure, recurrence, or death due to any cause.
  * Patients will be assessed for response according to modified International Working Group (IWG) criteria for MDS
Event-free survival in MDS patients treated with CPX-351 in patients undergoing allogeneic hematopoietic cell transplant | 1 year
  * Defined as the interval from the date of first dose of study drug to date of treatment failure, recurrence, or death due to any cause.
  * Patients will be assessed for response according to modified International Working Group (IWG) criteria for MDS

CONTACTS AND LOCATIONS:
Overall Officials: Meagan Jacoby, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu